CLINICAL TRIAL: NCT03002545
Title: Effects of a 12-week Supplementation With 400 mg Magnesium From Magnesium Citrate on Blood Sugar, Blood Pressure and Expression of Magnesium-sensitive Genes in Patients With Type II Diabetes
Brief Title: Magnesium Supplementation in Type II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Protina Pharmazeutische GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DiaMag 2017
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Effect of Magnesium in Diabetes
Keywords: Magnesium; Type II diabetes; magnesium-sensitive genes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): identically tasting and looking Placebo
  Interventions: Dietary Supplement: Placebo
- Magnesium (Active Comparator): Supplementation with 400 mg Magnesium from Magnesium citrate once daily
  Interventions: Dietary Supplement: Magnesium citrate

INTERVENTIONS:
Dietary Supplement: Magnesium citrate
  Arms: Magnesium
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This study aims to determine how a 12-week magnesium supplementation with 400 mg magnesium from organic magnesium citrate affects blood glucose control and insulin resistance within patients with type 2 diabetes (HbA1c> 6%) and how the expression of certain Mg-sensitive transporting genes is affected .

DETAILED DESCRIPTION:
The examinations are carried out in 50 subjects aged 20-80 years with existing type 2 diabetes (HbA1c> 6%). The target parameters are determined in the blood. Blood sampling takes place at confinement, after 6 weeks and at the end of the study (week 12). In addition, blood pressure is determined and general health condition of each subject is recorded by a standardized questionnaire (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Type II Diabetics (HbA1c > 6%)

Exclusion Criteria:

* pregnancy, lactation
* persons with severe renal impairment (glomerular filtration rate <30 ml / min)
* use of insulin, oral antidiabetic drugs, diuretics, antacids or proton pump inhibitors within 4 weeks prior to study start and during the study
* intake of vitamin supplements, dietary supplements, mineral products or possibly enriched foods containing Magnesium within 4 weeks before study start and during the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12; Primary Completion 2019-03 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
blood sampling | 12 weeks
  measurement of type II Diabetes relevant Parameters including Glucose, HbA1c, HOMA-IR, magnesium-sensitive gene expression
blood pressure measurement | 12 weeks
  measurement of blood pressure
questionnaire SF-36 | 12 weeks
  questionnaire is used to assess the physiological health Status of patients

CONTACTS AND LOCATIONS:
Locations (1):
- St. Anna Hospital, Herne, Germany